CLINICAL TRIAL: NCT02109367
Title: Diagnostic Utility of Culdocentesis in Patients With a Suspicious Adnexal Mass
Status: Active, not recruiting | Type: Observational
Sponsor: Southern Illinois University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BRARD-SIUSOM-14-001; 1R03CA181907-01 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; ovarian mass; CA-125; HE4; culdocentesis; biomarker(s)
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fluid sample infused and collected from the cul-de-sac
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic mass: Women who present to the Gynecologic Oncology clinic with a pelvic mass who are scheduled to undergo surgical excision.

SUMMARY:
This study involves women who are scheduled to have surgery for a pelvic or ovarian mass that is suspicious for epithelial ovarian cancer (EOC). The physician will perform an additional procedure on all consented subjects known as 'culdocentesis'. This will be done just prior to their scheduled surgery while the patient is under general anesthesia. Culdocentesis is a procedure typically used to check for abnormal fluid in the space just behind the vagina. This pocket of space is called the cul-de-sac. The purpose of this study is to determine if levels of tumor markers, CA-125 and HE4, are measurable from the cul-de-sac fluid. If these tumor markers are measurable from the cul-de-sac fluid and correlate with the patient's diagnosis, this procedure may be used in the future as an additional diagnostic tool for EOC. In addition, a single urine sample will be collected from each patient to measure the ratio of "good" to "bad" estrogen. Investigators hypothesize this ratio will also correlate with EOC diagnosis. Study results could lead to development of an alternative, minimally invasive and low risk diagnostic tool in patients with an ovarian mass suspicious for malignancy.

DETAILED DESCRIPTION:
This is a single cohort, exploratory pilot study of 60 participants to assess if ovarian cancer markers, cancer antigen-125 (CA-125) and human epididymis protein 4 (HE4), are measurable from cul-de-sac washings collected via culdocentesis. Immediately prior to the scheduled surgery, while the patient is under general anesthesia, a long, thin needle will be inserted through the wall of the vagina (just below the uterus) to access the cul-de-sac. A saline wash will then be performed and this fluid will be collected for analysis of tumor markers. CA-125 and HE4 levels will be compared to serum levels for correlation with a diagnosis of ovarian cancer. A urine sample will also be collected from this same cohort to measure estrogen metabolites. Estrogen metabolism is associated with cancer progression in estrogen sensitive tissues. Estrogen metabolites, 2-hydroxyestrone (2-OHE1) the "good" byproduct and 16α-hydroxyestrone (16α-OHE1) known as the "bad" byproduct, have been implicated in the development of breast cancer. Study investigators are proposing to expand the utility of this predictive ratio to ovarian cancer by measuring the potential imbalance of these metabolites.

If results indicate an association between cancer diagnosis and levels of CA-125 and HE4 or the ratio of estrogen metabolites from the urine, this could allow for a new minimally invasive, low-risk diagnostic modality for all suspected ovarian cancer cases. This would be particularly invaluable for patients at higher risk for poor surgical outcomes. Data from this pilot study will confirm the potential effect size needed to identify an optimal cut-point useful for the prediction of EOC within this study population.

ELIGIBILITY:
Inclusion criteria:

* Patients age ≥ 30.
* Adnexal mass or suspected ovarian carcinoma.
* Patient has been scheduled for oophorectomy, bilateral salpingo- oophorectomy (BSO), hysterectomy, hysterectomy/BSO, staging or debulking.
* Willingness to sign an Informed Consent document.

Exclusion criteria:

* Patients previously diagnosed with a malignancy within the pelvis or abdomen.
* Patients in which culdocentesis is technically unfeasible due to previous surgery (extensive pelvic floor repair/colpocleisis) or other anatomic abnormalities that make the cul-de-sac inaccessible.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women with a suspicious adnexal mass that could possibly be ovarian cancer who are scheduled for oophorectomy, bilateral salpingo-oophorectomy (BSO), hysterectomy via laparotomy or laparoscopy, hysterectomy/BSO, staging and/or debulking.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
HE4 and CA-125 from cul-de-sac wash | baseline
  ELISA

SECONDARY OUTCOMES:
2-hydroxyestrone (2-OHE1) and 16α-hydroxyestrone (16α-OHE1) from urine | baseline
  ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brard, MD, PhD, Principal Investigator — Southern Illinois University
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen MR, Goff BA, Lowe KA, Scholler N, Bergan L, Drescher CW, Paley P, Urban N. Use of a Symptom Index, CA125, and HE4 to predict ovarian cancer. Gynecol Oncol. 2010 Mar;116(3):378-83. doi: 10.1016/j.ygyno.2009.10.087. Epub 2009 Nov 28. PMID 19945742
- [Background] Bast RC Jr. Status of tumor markers in ovarian cancer screening. J Clin Oncol. 2003 May 15;21(10 Suppl):200s-205s. doi: 10.1200/JCO.2003.01.068. PMID 12743135
- [Background] Moore RG, Brown AK, Miller MC, Skates S, Allard WJ, Verch T, Steinhoff M, Messerlian G, DiSilvestro P, Granai CO, Bast RC Jr. The use of multiple novel tumor biomarkers for the detection of ovarian carcinoma in patients with a pelvic mass. Gynecol Oncol. 2008 Feb;108(2):402-8. doi: 10.1016/j.ygyno.2007.10.017. Epub 2007 Dec 3. PMID 18061248
- [Background] Partheen K, Kristjansdottir B, Sundfeldt K. Evaluation of ovarian cancer biomarkers HE4 and CA-125 in women presenting with a suspicious cystic ovarian mass. J Gynecol Oncol. 2011 Dec;22(4):244-52. doi: 10.3802/jgo.2011.22.4.244. Epub 2011 Dec 5. PMID 22247801
- [Background] Sandri MT, Bottari F, Franchi D, Boveri S, Candiani M, Ronzoni S, Peiretti M, Radice D, Passerini R, Sideri M. Comparison of HE4, CA125 and ROMA algorithm in women with a pelvic mass: correlation with pathological outcome. Gynecol Oncol. 2013 Feb;128(2):233-8. doi: 10.1016/j.ygyno.2012.11.026. Epub 2012 Nov 28. PMID 23200911